CLINICAL TRIAL: NCT01663012
Title: A Phase II, Single Arm, Open Label Study Of NKTR-102 In Bevacizumab-Resistant High Grade Glioma
Brief Title: Phase II NKTR-102 In Bevacizumab-Resistant High Grade Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lawrence Recht (Other)
Collaborators: Nektar Therapeutics (Industry)
Responsible Party: Sponsor-Investigator, Lawrence Recht, Professor of Neurology and Neurological Sciences, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-24833; SU-06212012-10228 (Other: Stanford University); NCI-2012-01288 (Other: National Cancer Institute); BRN0021 (Other: OnCore)
Record Dates: First submitted 2012-08-02; First posted 2012-08-13 (Estimated); Results first posted 2015-06-11 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-01

CONDITIONS: Anaplastic Astrocytomas; Anaplastic Oligodendrogliomas; Glioblastomas (GBM)
MeSH Terms: conditions — Astrocytoma; Oligodendroglioma; Glioblastoma | interventions — etirinotecan pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Drug: Etirinotecan pegol (Experimental): 145 mg/m2 dose
  Interventions: Drug: Etirinotecan pegol

INTERVENTIONS:
Drug: Etirinotecan pegol
  Other Names: NKTR-102

SUMMARY:
High Grade Gliomas, including anaplastic astrocytomas, anaplastic oligodendrogliomas and glioblastomas (GBM), are the most common and most aggressive primary brain tumors. Prognosis for patients with high-grade gliomas remains poor. The estimated median survival for patients with GBM is between 12 to 18 months. Recurrence after initial therapy with temozolomide and radiation is nearly universal. Since May 2009, the majority of patients in the US with an initial recurrence of high-grade glioma receive bevacizumab, a monoclonal antibody against vascular endothelial growth factor (VEGF), which is thought to prevent angiogenesis in these highly vascular tumors. BEV has response rates from 32-62% and has improved overall median survival in patients with recurrent high-grade gliomas1. However, the response is short lived, and nearly 100% of patients eventually progress despite bevacizumab. No chemotherapeutic agent administered following progression through bevacizumab has made a significant impact on survival. Patients progress to death within 1-5 months after resistance develops. Therefore, patients with high-grade gliomas who have progressed through bevacizumab represent a population in dire need of a feasible and tolerable treatment.

NKTR-102 is a topoisomerase I inhibitor polymer conjugate that was engineered by attaching irinotecan molecules to a polyethylene glycol (PEG) polymer using a biodegradable linker. Irinotecan released from NKTR-102 following administration is further metabolized to the active metabolite, 7-ethyl-10-hydroxy-camptothecin (SN38), that causes DNA damage through inhibition of topoisomerase. The goal in designing NKTR-102 was to attenuate or eliminate some of the limiting side effects of irinotecan while improving efficacy by modifying the distribution of the agent within the body. The size and structure of NKTR-102 results in marked alteration in pharmacokinetic (PK) profile for the SN38 derived from NKTR-102 compared to that following irinotecan: the maximal plasma concentration (Cmax) is reduced 5- to 10-fold and the half-life (t1/2 ) of SN38 is increased from 2 days to approximately 50 days. This altered profile leads to constant exposure of the tumor to the active drug. In addition, the large NKTR-102 molecule does not freely pass out of intact vasculature, which may account for relatively higher concentrations of the compound and the active metabolites in tumor tissues in in vivo models, where the local vasculature may be relatively more permeable. A 145 mg/m2 dose of NKTR-102, the dose intended for use in this phase II clinical trial (and being used in the phase III clinical program), results in approximately the same plasma exposure to SN38 as a 350 mg/m2 dose of irinotecan, but exposure is protracted, resulting in continuous exposure between dosing cycles and lower Cmax. NKTR-102 was therefore developed as a new chemotherapeutic agent that may improve the clinical outcomes of patients.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven high-grade glioma (WHO III or IV) with astrocytic component and must be in recurrence after treatment with bevacizumab
* Patients must have received conventional radiation therapy of total radiation dosage (ranging from 5400 to 6000 cGy administered in daily fractions of 150 to 200 cGy over 6 weeks) with concurrent temozolomide.

Patients must have received bevacizumab and be in recurrence after bevacizumab treatment.

* Patients must be at least 28 days from last administration of cytotoxic chemotherapy and at least 14 days from the last administration of bevacizumab.

  * Patients must be >18 years of age.
  * Patients must have a life expectancy > 6 weeks
  * Patients must have a Karnofsky Performance Score (KPS) >=50
  * If female, patients of childbearing potential must have a negative serum beta-hCG pregnancy test and must agree to use hormonal or barrier birth control with spermicidal gel to avoid pregnancy during the study
  * Adequate organ function (obtained within 14 days prior to randomization and analyzed by the central laboratory) as evidenced by:

    1. Absolute neutrophil count (ANC) >=1.5 X 10^9/L without myeloid growth factor support for 7 days preceding the lab assessment;
    2. Hemoglobin (Hgb) >= 9 g/dL (90 g/L); < 9 g/dL (< 90 g/L) is acceptable if hemoglobin is corrected to >= 9 g/dL (90 g/L) as by growth factor or transfusion prior to randomization;
    3. Platelet count >=100 X 10^9/L without blood transfusions for 7 days preceding the lab assessment;
    4. Bilirubin <= 1.5 X upper limit of normal (ULN), except for patients with documented history of Gilbert's disease;
    5. Alanine aminotransferase (ALT), and aspartate aminotransferase (AST) <= 2.5 X ULN
    6. Alkaline phosphatase (AP) <= 3 X ULN
    7. Serum creatinine <= 1.5 mg/dL (133 µmol/L) or calculated creatinine clearance >= 50 mL/min (using Cockcroft-Gault formula);
    8. Women of childbearing potential (WCBP): negative serum pregnancy test (this test is required of all women unless post-menopausal, defined as 12 consecutive months since last regular menses, or surgically sterile).
  * Patients must be willing and able to comply with the protocol and provide written informed consent prior to study-specific screening procedures.

Exclusion Criteria:

Patients who meet any of the following criteria must not be permitted entry to the study.

* Patients who have had chemotherapy within 28 days, radiotherapy within 28 days, biological therapy within 14 days, and investigational therapy within 21 days prior to first dose of experimental drug.
* Patients who have received prior treatment for cancer with a camptothecin derivative (eg, irinotecan, topotecan, and investigational agents including but not limited to exatecan, rubitecan, gimatecan, karenitecan, SN38 investigational agents, EZN-2208, SN-2310, and AR-67).
* Patients with the following co-morbid disease or incurrent illness:

  1. Patients with chronic or acute GI disorders resulting in diarrhea of any severity grade; patients who are using chronic anti-diarrheal supportive care (more than 3 days/week) to control diarrhea in the 28 days prior to first dose of investigational drug.
  2. Patients with known cirrhosis diagnosed with Child-Pugh Class A or higher liver disease.
  3. Prior malignancy except for non-melanoma skin cancer and carcinoma in situ (of the cervix or bladder), unless diagnosed and definitively treated more than 3 years prior to first dose of investigational drug.
  4. Severe/uncontrolled inter-current illness within the previous 28 days prior to first dose of investigational drug.
  5. Significant known cardiovascular impairment (NYHA CHF > grade 2, unstable angina, myocardial infarction within the previous 6 months prior to first dose of investigational drug, or existing serious cardiac arrhythmia).
  6. Patients who require daily use of oxygen supplementation in the 28 days prior to first dose of investigational drug.
  7. Any other significant co-morbid conditions that in the opinion of the Investigator would impair study participation or cooperation.
* Patients with a known allergy or hypersensitivity to any of the components of the investigational therapy, including PEG or topoisomerase inhibitors.
* Patients receiving the following medications at the time of first dose of investigational drug:

  * Pharmacotherapy for hepatitis B or C, tuberculosis, or HIV.
  * enzyme inducing anti-epileptic medications (EIAEDs)
  * other chemotherapy, other investigational agents , or biologic agents for
  * the treatment of cancer including antibodies(eg, bevacizumab,
  * trastuzumab, or pertuzumab) or any investigational agent(s).
* Pregnant or nursing patients will be excluded from the study.
* Patients receiving active treatment for HIV will be excluded from this study because non-nucleoside reverse transcriptase inhibitors, protease inhibitors and maraviroc (a CCR5-antagonist) are extensively metabolized by the cytochrome P450 system. Interactions with these drugs may induce or inhibit irinotecan or SN38 metabolism, leading to over or under-dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-07; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Recht, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Palo Alto, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Drug: Etirinotecan Pegol: 145 mg/m2 dose
  Etirinotecan pegol
Period: Overall Study
Arm/Group | Drug: Etirinotecan Pegol
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Drug: Etirinotecan Pegol
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 3
Age, Continuous [Median (Full Range); unit: years] | 49.5 [20 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival, Assessed by Revised Assessment in Neuro-oncology (RANO) Criteria
Description: Will be described using Kaplan-Meier estimates. The PFS probability at 6 weeks (PFS-6week) will be estimated with an 80% power and 95% confidence intervals (80% in accord with the planned alpha level, 95% for comparability with other studies, confidence intervals based on the Greenwood formula for the variance of a survival probability).
Time Frame: 6 weeks from first administration of NKTR-102
Measure: Number; unit: participants
Arm/Group | Drug: Etirinotecan Pegol
Number analyzed (Participants) | 20
participants | 11

2. Secondary Outcome: Survival From the Time of First NKTR-102 Dose for Patients With BEV-resistant Glioma Receiving NKTR-102 to Date of Death
Description: Will be described using Kaplan-Meier estimates.
Time Frame: From date of first dose of NKTR-102 to date of death, assessed up to 2 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Drug: Etirinotecan Pegol
Number analyzed (Participants) | 20
Months | 4.5 [2.4 to 5.9]

3. Secondary Outcome: Overall Survival From Time of Diagnosis
Description: Will be described using Kaplan-Meier estimates.
Time Frame: From date of pathologic diagnosis/confirmation of high grade glioma to date of death, assessed up to 2 years.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Drug: Etirinotecan Pegol
Number analyzed (Participants) | 20
Months | 17.1 [10.0 to 36.6]

ADVERSE EVENTS:
Time Frame: Open-ended until 30 days after last dose of Etirinotecan Pegol
Arm/Group | Drug: Etirinotecan Pegol
Serious Adverse Events (participants affected / at risk) | 5/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug: Etirinotecan Pegol (N=20)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dehyrdation (Metabolism and nutrition disorders) | 1 (2)
Hyponatermia (Metabolism and nutrition disorders) | 1 (1)
Malignant Neoplasms, Brain Primary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 2 (2)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug: Etirinotecan Pegol (N=20)
Neutrophil Count Decreased (Blood and lymphatic system disorders) | 3 (4)
Palpitations (Cardiac disorders) | 1 (2)
Blurred Vision (Eye disorders) | 9 (13)
Dry Eye (Eye disorders) | 1 (1)
Eye Twitching (Eye disorders) | 2 (2)
Pressure Behind Eyes (Eye disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 5 (7)
Constipation (Gastrointestinal disorders) | 8 (8)
Diarrhea (Gastrointestinal disorders) | 14 (41)
Fecal Incontinence (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 2 (3)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 4 (5)
Tongue Swelling (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 14 (21)
Toothache (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 9 (9)
Edema Limbs (General disorders) | 2 (2)
Fatigue (General disorders) | 12 (18)
Non Cardiac Chest Pain (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Bladder Infection (Infections and infestations) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 2 (5)
Fall (Injury, poisoning and procedural complications) | 1 (4)
Alanine Aminotransferase Increased (Investigations) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 6 (7)
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Left Sided Muscle Weakness (Musculoskeletal and connective tissue disorders) | 2 (3)
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 2 (3)
Cognative Disturbance (Nervous system disorders) | 2 (3)
Dizziness (Nervous system disorders) | 6 (7)
Dysphasia (Nervous system disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 7 (11)
Peripheral Motor Neuropathy (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 8 (11)
Somnolence (Nervous system disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1)
Bladder Spasm (Renal and urinary disorders) | 1 (1)
Urinary Incontinence (Renal and urinary disorders) | 2 (2)
Urinary Tract Pain (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No